CLINICAL TRIAL: NCT06727175
Title: A Multi-center Efficacy Study of Noninvasive Neuromodulation in the Treatment of Subjective Tinnitus
Brief Title: A Multicenter Study of Noninvasive Neuromodulation Treatment for Subjective Tinnitus
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-671-01
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Subjective Tinnitus
Keywords: non-invasive neuromodulation; Subjective tinnitus; clinical effect; sleep quality; anxiety; depression
MeSH Terms: conditions — Tinnitus; Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- before non-invasive neuromodulation therapy: evaluation results before non-invasive neuroregulation therapy
  Interventions: Other: before any intervention
- after non-invasive neuromodulation therapy: evaluation results after six-month non-invasive neuroregulation therapy
  Interventions: Behavioral: non-invasive neuromodulation therapy

INTERVENTIONS:
Behavioral: non-invasive neuromodulation therapy — Patients with subjective tinnitus were treated using non-invasive neuroregulation therapy. That is, to generate personalized, non-invasive acoustically stimulated neuroregulation regimens for six montns. Each participant was treated three times a day (morning, noon and bedtime) for 30 minutes each time.
  Groups: after non-invasive neuromodulation therapy
Other: before any intervention — before any intervention
  Groups: before non-invasive neuromodulation therapy

SUMMARY:
The purpose of this study is to find out the scientific and effectiveness of non-invasive neuromodulation therapy for subjective tinnitus and further guide the clinical response to tinnitus problems. This study collects the case data of subjective tinnitus patients who received non-invasive neuromodulation treatment for statistical analysis. The complete data included pure tone audiometry, tinnitus assessment, mood assessments, and sleep quality assessment. Paired T-tests are suppoesed to be conducted to analyze the clinical efficacy of non-invasive neuromodulation therapy for subjective tinnitus and its specific effect on improving mood and sleep.

DETAILED DESCRIPTION:
The purpose of this study is to find out the scientific and effectiveness of non-invasive neuromodulation therapy for subjective tinnitus and further guide the clinical response to tinnitus problems. This study collects the case data of subjective tinnitus patients who received non-invasive neuromodulation treatment for statistical analysis. The complete data included pure tone audiometry, tinnitus assessment (tinnitus matching, Tinnitus Handicap Inventory, Tinnitus Function Index, Visual analog Scales), mood assessments (Hamilton Anxiety Scale, Hamilton Depression Scale), and sleep quality assessment (Pittsburgh Sleep Index Scale). Paired T-tests are suppoesed to be conducted to analyze the clinical efficacy of non-invasive neuromodulation therapy for subjective tinnitus and its specific effect on improving mood and sleep.

ELIGIBILITY:
Inclusion Criteria:

* ≥18yrs,
* Diagnosed as subjective tinnitus,
* THI≥38,
* Chinese, can cooperate with all Chinese version evaluation,
* Right-handed,
* No major neurological disease or other

Exclusion Criteria:

* Hyperacustic,
* Incomplete case data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjective tinnitus patients and compliance with 6 months of noninvasive neuromodulation therapy, with complete two-assessment scale records.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
tinnitus loudness | 0-7 days pre-therapy, 0-7 days post-therapy
  Taking 1dB as the step, parrticipants were asked to select the signal sound intensity consistent with their subjective tinnitus loudness, and the tinnitus loudness matching was completed after repeated testing. The difference between the matched intensity and the pure tone hearing threshold at this frequency was recorded as tinnitus loudness (dB SL).
tinnitus handicap inventory, THI | 0-7 days pre-therapy, 0-7 days post-therapy
  THI is divided into three sub-scales, namely functional, emotional and catastrophic. THI contains a total of 25 items, and each item is scored 4, 2 and 0 points according to "yes", "sometimes" and "no" respectively. After each item score was completed, the THI total score, THI functional total score (THI-F), THI affective total score (THI-E), and THI catastrophic total score (THI-C) were calculated for the specific patient. The severity of tinnitus was evaluated according to the total score: 1-16 points, grade 1 (slight); 18-36 points, grade 2 (mild); 38-56pointks, grade 3 (moderate); 58-76 points, level 4 (severe); Score 78-100, level 5 (catastrophic).
tinnitus functional index, TFI | 0-7 days pre-therapy, 0-7 days post-therapy
  The scale contains 8 subscales. They are denoted as TFI-I (Intrusiveness) and TFI-SC (Sense of) control), TFI-C (Cognition), TFI-S (Sleep), TFI-A (Auditory), TFI-R (Relaxation), TFI-Q (Quality of life), TFI-E (Emotional) distress); A total of 25 items are included. Each item is worth 100 points. The average score of all items is recorded as the total TFI score. The higher the score, the higher the pain and severity of the subject's tinnitus.
visual analogue scale, VAS | 0-7 days pre-therapy, 0-7 days post-therapy
  VAS was used to evaluate the impact of tinnitus on the daily life of patients with chronic subjective tinnitus. Scale 0-10. A score of 0 means that tinnitus has no impact on daily life, and a score of 10 means that tinnitus has an intolerable, fatal level of impact on daily life. VAS was used to evaluate subjective tinnitus loudness, annoyance, depression, and tinnitus control difficulty.

SECONDARY OUTCOMES:
Hamilton Anxiety Scale, HAMA | 0-7 days pre-therapy, 0-7 days post-therapy
  The scale contains 14 items, mainly involving two aspects of physical anxiety and mental anxiety. The scale is scored on a 0-4 scale on five scales: 0 for asymptomatic, 1 for mild, 2 for moderate, 3 for severe, and 4 for extremely severe.
Hamilton depression scale, HAMD | 0-7 days pre-therapy, 0-7 days post-therapy
  The study uses a 24-item version. Each item is scored on a 0-4 scale on a 5-point scale: 0 for asymptomatic, 1 for mild, 2 for moderate, 3 for severe, and 4 for extremely severe.
Pittsburgh sleep quality index, PSQI | 0-7 days pre-therapy, 0-7 days post-therapy
  The scale contains 24 items, which are divided into subjective sleep quality, sleep time, sleep latency, sleep efficiency, sleep disorders, sleep medication use and daily dysfunction, with a total of 7 components. Each component is rated 0-3 points. The total score ranges from 0 to 21. The higher the score, the worse the sleep quality in the past month. Among them, 0-5 points represent excellent sleep quality, 6-10 points represent good sleep quality, 11-15 points represent moderate sleep quality, 16-20 points indicate poor sleep quality, and 21 points indicate the worst sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Haidi Yang, PhD, Study Director — SunYatSunU2H
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong 510000, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No